CLINICAL TRIAL: NCT01426750
Title: Enteral Nutrition Support in Children and Adolescents With Cancer: a Non-randomized Controlled Clinical Trial
Brief Title: Enteral Nutrition Support in Children and Adolescents With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPM 1463/7
Record Dates: First submitted 2008-03-28; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Malnutrition; Cancer
Keywords: Nutritional support.; Cancer.; Malnutrition.; Child.; Adolescent
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IOS, TFR (Experimental): industrialized oral supplementation (IOS) and tube feeding regimen (TFR) with Nutren 1.0 or Jr (Nestlé-Clinical Nutrition).
  Interventions: Dietary Supplement: industrialized oral supplementation (IOS) and tube feeding regimen (TFR) with Nutren

INTERVENTIONS:
Dietary Supplement: industrialized oral supplementation (IOS) and tube feeding regimen (TFR) with Nutren — The oral and tube supplement offered was Nutren Jr® (for patients aged 1 - 9 years) or Nutren 1.0- Nestlé Clinical Nutrition-Brazil (for those aged 10 years or over). This supplement was a whole powder formulation that presented a macro composition of 52% carbohydrates, 12% proteins and 36% lipids. Its vitamins were A, D, E, K, B complex, biotin and choline; its trace elements were iron, copper, zinc, manganese, selenium, chromium and molybdenum; its macroelements were potassium, calcium, sodium, chlorine, iodine, magnesium and phosphorus; and it contained taurine and L-carnitine presenting 1.0 kcal/ml.

SUMMARY:
CONTEXT AND OBJECTIVE: Tumor and its therapy have adverse effects on the nutritional status of cancer patients, leading to nutritional support. The aim was to study enteral nutrition indications, as well as its compliance and the impact on nutritional status.

DESIGN AND SETTING: Clinical trial, IOP, Unifesp-EPM. METHODS: Patients older than 1 year followed during anticancer therapy were included from January 2002 to January 2004. They received industrialized oral supplementation - Nutren 1.0 or Jr (IOS) and were followed on a weekly basis and reevaluated on weeks 3, 8 and 12: at these times, if inadequate outcome was observed, tube feeding with the same supplement (TFR) was indicated.

ELIGIBILITY:
Inclusion Criteria:

* Were chemotherapy, age above one year and malnutrition
* A z-score of weight for height (zW/H) < -1.0 to -2.0 in children26 and ≥ 5th to < 15th of body mass index (BMI) in adolescents 27 were considered as mild malnutrition
* A zW/H < -2.0 in children and < 5th of BMI in adolescents as severe, respectively.28 In adults, the World Health Organization (WHO)29 cut-off values were applied: < 18.5 mild and < 17 severe malnutrition.

Exclusion Criteria:

* Were corticosteroid or hormonal therapy
* Swallowing abnormalities
* Parenteral or tube feeding therapy
* Palliative care and presence of non cancer-related diseases.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)